CLINICAL TRIAL: NCT04514913
Title: Study of Focal Airway Disease in Asthma Using Image Guided Bronchoscopy
Acronym: SOFA
Status: Withdrawn | Type: Observational
Why Stopped: The restrictions on research imposed for the COVID-19 pandemic prevented us from launching study recruitment and visits. At this stage our funding is not sufficient to allow us to enroll sufficient numbers of patients so we will close the study.
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-27331; 2P01HL107202-06A1 (NIH)
Record Dates: First submitted 2020-08-12; First posted 2020-08-17 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Asthma; Mucus; Plug, Tracheobronchial
Keywords: Asthma; Mucus Plug; Bronchoscopy; CT Scan
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — bronchoalveolar lavage from airways in 1-2 bronchopulmonary segments, bronchial brushes from airways in 2-3 bronchopulmonary segments, endobronchial biopsies from airways in 2-3 bronchopulmonary segments, and blood.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Controls: Participants with no history of asthma or other lung diseases.
  Interventions: Radiation: Multidetector Computed Tomography (MDCT) Scan; Procedure: Virtual Navigation Bronchoscopy (VNB)
- Asthmatics without mucus plugs: Participants with asthma and no evidence of mucus plugging.
  Interventions: Radiation: Multidetector Computed Tomography (MDCT) Scan; Procedure: Virtual Navigation Bronchoscopy (VNB)
- Asthmatics with mucus plugs: Participants with asthma and evidence by MDCT lung scan showing mucus plugging.
  Interventions: Radiation: Multidetector Computed Tomography (MDCT) Scan; Procedure: Virtual Navigation Bronchoscopy (VNB)

INTERVENTIONS:
Radiation: Multidetector Computed Tomography (MDCT) Scan — This is a low-dose CT scan of the chest using no contract material.
Procedure: Virtual Navigation Bronchoscopy (VNB) — This is a procedure where a camera will be inserted into the lung in order to guide sample collection of bronchoalveolar lavages, bronchail brushes and endobronchial biopsies.

SUMMARY:
This is a single center study of 60 subjects including those with asthma and mucus plugging, those with asthma and without mucus plugging, and healthy controls. Screening data will be reviewed to determine participant eligibility. Participants who meet all inclusion criteria will participate in image-guided bronchoscopy ("virtual navigation bronchoscopy" [VNB]) to sample airway biospecimens in mucus plugged and control airways.

DETAILED DESCRIPTION:
This is a single center study of 60 subjects. The investigators will enroll 30 subjects with asthma who demonstrate mucus plugging on a screening CT lung scan, 15 subjects with asthma without mucus plugging, and 15 healthy controls. The healthy controls and subjects with asthma but without mucus plugging with also undergo CT scans to confirm that their lungs aren't obstructed by mucus.

Screening data will be reviewed to determine participant eligibility. Participants who meet all inclusion criteria will participate in image-guided bronchoscopy ("virtual navigation bronchoscopy" [VNB]) to sample airway biospecimens in mucus plugged and control airways. Subjects will participate in up to 5 study visits at the Airway Clinical Research Center.

ELIGIBILITY:
Group 1: Healthy Controls

Inclusion Criteria:

* Male or female between the ages of 18 and 70 years at Visit 1 and at least 50% whose age is > 40 years (to ensure age balance among groups and anticipating that group 3 subjects will be older).
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
* Able to perform reproducible spirometry according to ATS criteria.

Exclusion Criteria:

* Upper respiratory tract infection (URI) within the previous 6 weeks.
* History of lung disease.
* Smoking of tobacco or other recreational inhalants in last month and/or >10 pack-year smoking history.
* Currently pregnant.
* History of allergic rhinitis.
* Laboratory evidence of atopy (blood eosinophils > 0.4 cells/dL, IgE > 165 IU/mL)
* History of unstable cardiovascular disease.
* BMI > 45
* Currently taking anticoagulants.

Group 2: Asthmatic Subjects without Mucus Plugs

Inclusion Criteria:

* Male or female between the ages of 18 and 70 years at Visit 1 and at least 50% whose age is > 40 years (to ensure age balance among groups and anticipating that group 3 subjects will be older).
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
* Able to perform reproducible spirometry according to ATS criteria.
* Physiological evidence of airflow obstruction (FEV1 bronchodilator reversibility of ≥ 12% or hyperreactivity to methacholine reflected by a methacholine PC20 ≤ 16 mg/mL). Historical methacholine data from previous studies conducted in the past 5 years at the UCSF ACRC will be allowed.
* Clinical history of asthma per patient report or medical record.
* Asthma requiring treatment with inhaled corticosteroids (ICS) for 3 months or greater.

Exclusion Criteria:

* Asthma exacerbation or URI within the previous 6 weeks.
* Currently pregnant.
* Smoking of tobacco or other recreational inhalants in last month and/or >10 pack-year smoking history.
* Other chronic pulmonary disorders, including cystic fibrosis and chronic obstructive pulmonary disease.
* History of unstable cardiovascular disease.
* BMI > 45.
* Currently taking anticoagulants.

Group 3: Asthmatic Subjects with Mucus Plugs

Inclusion:

* Male or female between the ages of 18 and 70 years at Visit 1.
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
* Able to perform reproducible spirometry according to ATS criteria.
* Physiological evidence of airflow obstruction (FEV1 bronchodilator reversibility of ≥ 12% or hyperreactivity to methacholine reflected by a methacholine PC20 ≤ 16 mg/mL). Historical methacholine data from previous studies conducted in the past 5 years at the UCSF ACRC will be allowed.
* Clinical history of asthma per patient report or medical record.
* Asthma requiring treatment with inhaled corticosteroids (ICS) for 3 months or greater.
* A MDCT lung scan indicating a mucus plug accessible by bronchoscopy in at least one airway.

Exclusion Criteria:

* Asthma exacerbation or URI within the previous 6 weeks.
* Currently pregnant.
* Smoking of tobacco or other recreational inhalants in last month and/or >10 pack-year smoking history.
* Other chronic pulmonary disorders, including cystic fibrosis and chronic obstructive pulmonary disease.
* History of unstable cardiovascular disease.
* BMI > 45.
* Currently taking anticoagulants.
* Mucus plugs inaccessible by bronchoscope.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with asthma who present with or without mucus plugs, as well as healthy controls, all between the ages of 18 and 70.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Difference in eosinophil percentage in broncheoalveolar biospecimens between asthmatic and non-asthmatic airways | 6 months
  The investigators will examine differences in type-2 inflammatory markers in bronchoalveolar biospecimens. Eosinophils are an indicator of type 2 inflammation in bronchial lavage samples. Indicators of airway inflammation will be compared with healthy control biospecimens and those of non-mucus plugged asthmatics.
Difference in gene expression of genes that mark IL-13 activation between asthmatic and non-asthmatic airways | 6 months
  Genes such as periostin, CLCA1, and Serpin B2 will be analyzed for expression in epithelial cell brushings.

CONTACTS AND LOCATIONS:
Overall Officials: John Fahy, MD, MSc, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Airway Clinical Research Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.

REFERENCES:
- See also: Airway Clinical Research Center website — http://acrc.ucsf.edu